CLINICAL TRIAL: NCT03913481
Title: Acute Normovolemic Hemodilution in High-risk Cardiac Surgery Patients. A Multicentre Randomized Trial.
Brief Title: Acute Normovolemic Hemodilution in High Risk Cardiac Surgery Patients.
Acronym: ANH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ANH/35/OSR
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: tissue; organ and systemic injury responses to surgery; trauma; burn; sepsis; hemorrhage; ischemia- reperfusion; resuscitation; including integrating pathways and signals; cardiac surgery; transfusion
MeSH Terms: conditions — Wounds and Injuries; Burns; Sepsis; Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANH (Experimental): Best available treatments plus ANH, performed withdrawing a volume of blood before the CPB. The volume will be personalized for every patient, but it'll be at least 650ml.
  Interventions: Procedure: Acute normovolemic hemodilution
- Standard care (Other): No ANH
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Acute normovolemic hemodilution — In the ANH arm, after induction of general anesthesia, a total blood volume of at least 650 ml of blood will be drawn from a central line. The amount of volume drawn can be replaced with Ringer lactate or a similar crystalloid fluid up to a 3:1 ratio.
  Arms: ANH
Procedure: Standard care — Best available treatment without ANH
  Arms: Standard care

SUMMARY:
Transfusions are one of the most overused treatments in modern medicine, and saving blood is one important issue all around the world. Cardiac surgery makes up a large percentage of the overall blood components consumption in surgery.

Acute normovolemic hemo-dilution (ANH) is a well-known strategy which has been used for years without the support of high quality evidence based medicine to improve post-cardiopulmonary bypass coagulation and reduce red blood cells (RBC) transfusion. We designed a multicenter randomized controlled trial to investigate the effect of ANH in reducing the number of cardiac surgery patients receiving RBC transfusions during hospital stay. We will randomize 2000 patients to have sufficient power to demonstrate a 20% relative and 7% absolute risk reduction in the number of patients' RBC transfusion. If the results of the study will confirm our hypothesis, this will have a great impact on blood management in cardiac operating room.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Any cardiac surgical intervention on CPB
* Elective surgery

Exclusion Criteria:

* Medical decision (e.g.: planned pre-CPB ANH considered undeniable for ethical reasons or not applicable for safety issues)
* Unstable Coronary Artery Disease: Recent (< 6 weeks) myocardial infarction, unstable angina, severe (> 70%) left main coronary artery stenosis
* Critical preoperative state (ventricular tachycardia or ventricular fibrillation or aborted sudden death, preoperative cardiac massage, preoperative ventilation before anesthetic room, hemodynamic instability, preoperative inotropes or IABP, preoperative severe acute renal failure (anuria or oliguria <10ml/hr.)
* Emergency surgery
* Pregnancy
* Unfeasibility to withdraw ≥ 650 ml without inducing hemodynamic instability
* Unfeasibility to withdraw ≥ 650 ml without inducing pre-CPB anemia (Htc <30%)
* Unfeasibility to withdraw ≥ 650 ml without inducing low Htc during CPB (Htc <24%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
RBCs transfusion | hospital discharge, an average of 10 days
  The number of patients receiving RBCs transfusion after elective cardiac surgery.

SECONDARY OUTCOMES:
Mortality | 30 days
  30-day mortality
Bleeding complications | hospital discharge, an average of 10 days
  * Amount of blood components (RBC, fresh frozen plasma-FFP, platelet -PLT) transfused (units/ml)
  * Estimated total blood volume lost (ml) at 12 hours after surgery
  * Surgical revision for bleeding
Ischemic complications | hospital discharge,an average of 10 days
  * Myocardial infarction
  * Stroke
  * Thromboembolic events
AKI | hospital discharge, an average of 10 days
  Developing of acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zangrillo, Prof, Study Chair — Vita-Salute University of Milano
Locations (32):
- United States (2):
  - OUHSC - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Virginia, Charlottesville, Virginia
- Mohammed Bin Khalifa Specialist Cardiac Center, Awali, Bahrain, Bahrain
- Brazil (2):
  - Dante Pazzanese Institute od Cardiology, São Paulo
  - Instituto do Coração - Hospital das Clínicas, Faculdade de Medicina - Universidade de São Paulo, São Paulo
- Xijing Hospital, Xi'an, China
- Italy (16):
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Azienda Ospedaliero Universitaria Policlinico "G.Rodolico - San Marco", Catania
  - Città di Lecce Hospital - GVM Care & Research, Lecce
  - IRCCS Policlinico San Donato, Milan
  - IRCCS Cardiologico Monzino, Milan
  - Ospedale San Raffaele di Milano, Italy, Milan
  - Azienda Ospedaliera Padova, Padua
  - AOU Pisana, Pisa
  - Ospedale San Carlo, Potenza
  - Policlinico Tor Vergata, Rome
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Rome
  - Istituto Clinico Humanitas, Rozzano
  - San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Russia (5):
  - Astrakhan Centre For Cardiac Surgery, Astrakhan
  - Moscow Clinical Scientific Center named after Loginov, Moscow
  - Vishnevsky National Medical Research Center of Surgery, Moscow
  - E. Meshalkin National Medical Research Center, Novosibirsk
  - Saint-Petersburg State University Hospital, Saint Petersburg
- King Abdullah Medical City, Mecca, Saudi Arabia
- Institute of Cardiovascular Diseases "Dedinje", Belgrade, Serbia
- National University Hospital, Singapore, Singapore
- Chiang Mai University Hospital, Chiang Mai, Thailand
- Kosuyolu High Specialization Education and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Monaco F, Guarracino F, Vendramin I, Lei C, Zhang H, Lomivorotov V, Osinsky R, Efremov S, Gurcu ME, Mazzeffi M, Pasyuga V, Kotani Y, Biondi-Zoccai G, D'Ascenzo F, Romagnoli E, Nigro Neto C, Do Nascimento VTNDS, Ti LK, Lorsomradee S, Farag A, Bukamal N, Brizzi G, Lobreglio R, Belletti A, Arangino C, Paternoster G, Bonizzoni MA, Tucciariello MT, Kroeller D, Di Prima AL, Mantovani LF, Ajello V, Gerli C, Porta S, Ferrod F, Giardina G, Santonocito C, Ranucci M, Lembo R, Pisano A, Morselli F, Nakhnoukh C, Oriani A, Pieri M, Scandroglio AM, Kirali K, Likhvantsev V, Longhini F, Yavorovskiy A, Bellomo R, Landoni G, Zangrillo A. Acute normovolemic hemodilution in cardiac surgery: Rationale and design of a multicenter randomized trial. Contemp Clin Trials. 2024 Aug;143:107605. doi: 10.1016/j.cct.2024.107605. Epub 2024 Jun 10. PMID 38866095
- [Background] Barile L, Fominskiy E, Di Tomasso N, Alpizar Castro LE, Landoni G, De Luca M, Bignami E, Sala A, Zangrillo A, Monaco F. Acute Normovolemic Hemodilution Reduces Allogeneic Red Blood Cell Transfusion in Cardiac Surgery: A Systematic Review and Meta-analysis of Randomized Trials. Anesth Analg. 2017 Mar;124(3):743-752. doi: 10.1213/ANE.0000000000001609. PMID 27669554
- [Derived] Monaco F, Lei C, Bonizzoni MA, Efremov S, Morselli F, Guarracino F, Giardina G, Arangino C, Pontillo D, Vitiello M, Belletti A, Ajello V, Licheri M, Nigro Neto C, Barucco G, Bukamal NA, Faustini C, Mantovani LF, Oriani A, Santonocito C, Mucchetti M, Federici F, Gerli C, Porta S, Scandroglio AM, Zhang H, Pieri M, Osinsky R, Lazzari S, Leonova E, Calabro MG, Amitrano D, Turi S, Prati P, Fresilli S, D'Amico F, D'Andria Ursoleo J, Labanca R, Marmiere M, Pruna A, Scquizzato T, Kirali K, Monti G, Carmona MJC, Tanaka K, Likhvantsev V, Ti LK, Bove T, Paternoster G, Singh K, Gurcu ME, Lomivorotov V, Landoni G, Bellomo R, Zangrillo A; ANH Study Group. A Randomized Trial of Acute Normovolemic Hemodilution in Cardiac Surgery. N Engl J Med. 2025 Jul 31;393(5):450-460. doi: 10.1056/NEJMoa2504948. Epub 2025 Jun 12. PMID 40503713